CLINICAL TRIAL: NCT04823325
Title: Use of Biomarkers in Early Surgery Patients to Determine Effectiveness of Regional Acceleratory Phenomenon and Its Effect on Root Resorption
Brief Title: Determining the Presence of RAP in Orthognathic Patients and Its Effect on Root Resorption by Biomarkers
Acronym: RAP
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: bkilic001
Record Dates: First submitted 2021-03-10; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Class III Malocclusion; Root Resorption
MeSH Terms: conditions — Malocclusion, Angle Class III; Root Resorption | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery patients: Otherwise healthy patients with Skeletal Class III problem
  Interventions: Procedure: Orthognathic Surgery

INTERVENTIONS:
Procedure: Orthognathic Surgery — The duration for presurgical orthodontic treatment was; 7,7 ± 1,7 months.

SUMMARY:
A prospective clinical trial to what extent inflammatory biomarkers are affected by the medication after orthognathic surgery in early surgical cases and whether these biomarkers affects the amount of maxillary or mandibular incisor root resorption.

DETAILED DESCRIPTION:
To conduct a prospective clinical trial to what extent inflammatory biomarkers such as OPG, RANKL, IL-1, IL-6, and CRP are affected by the medication after orthognathic surgery in early surgical cases and whether these biomarkers affects the amount of maxillary or mandibular incisor root resorption.

ELIGIBILITY:
Inclusion Criteria

1. Have skeletal Cl III malocclusion
2. Wisdom teeth are absent or extracted at least 6 months before the surgery
3. Need of orthognathic surgery through Le Fort I osteotomy of the maxilla and bilateral sagittal split osteotomies (BSSO) of the mandible.
4. Undergo fixed orthodontic treatment before and after the orthognathic surgery
5. Have available orthopantomograms with adequate quality
6. Have healthy periodontal tissue without inflammation or bleeding before and after the surgery.
7. Maintain the same medication protocol during and after the surgery.

Exclusion Criteria:

1. ongoing use of regular medication
2. smoking
3. known penicillin allergy,
4. any immune disorder,
5. musculoskeletal diseases,
6. syndromes,
7. cleft lip-palate,
8. systemic diseases affecting root resorption,
9. periodontal and gingival disorders,
10. missing teeth among upper or lower incisors,
11. poor oral hygiene.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study was started by collecting GCF before surgery from 25 patients. Patients who developed exclusion criteria while the study was in progress were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Assessing Change Between Three Time Points of Biomarkers to Determine Effectiveness of Regional Acceleratory Phenomenon | To see the change at biomarker levels GCF samples were collected at the time points designated as T0, T1, and T2 which correspond to the day of the surgery before anesthesia, 1 week after the surgery, and 4 weeks after the surgery
  IL- 6 RANKL
Assessing Change Between Two Time Points to Determine Root Resorption | To see the change of root length all radiographs were taken digitally at t0 (at the beginning of orthodontic preparation), t1 (just before the orthognathic surgery), and t2 ( an average of 1,5 years postop) with an X-ray unit
  Morphologic changes in root apex

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kilic, Study Director — Bezmialem Vakif University; Nisa Gül Amuk, Principal Investigator — TC Erciyes University
Locations (1):
- Banu Kilic, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No